CLINICAL TRIAL: NCT03149926
Title: Emotional Reaction of Patients With Borderline Personality Disorder (BPD)on Stimuli Connected to Self-injury - A Comparison Between Patients With BPD and a Healthy Control Group.
Brief Title: Emotional Reaction and Self Injury in Patients With Borderline Personality Disorder and Healthy Controls
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Katharina Bachmann (Other)
Responsible Party: Sponsor-Investigator, Katharina Bachmann, Psychologist Msc., University of Oldenburg
Organization: University of Oldenburg (Other)
Other Study IDs: UOldenburg2
Record Dates: First submitted 2017-05-09; First posted 2017-05-11 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Borderline Personality Disorder; Emotions
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Borderline Personality Disorder
  Interventions: Other: Stimuli presentation
- Healthy controls
  Interventions: Other: Stimuli presentation

INTERVENTIONS:
Other: Stimuli presentation — Different stimuli associated with self-injury are presented. Participants have to rate the emotional effect elected by the stimuli.

SUMMARY:
The current study investigates the emotional response of patients with borderline personality disorder and healthy controls on stimuli associated with self-injury.

ELIGIBILITY:
Inclusion Criteria:

* Patients that are able to use skills and have some therapy experiences.

Exclusion Criteria:

* Severe psychiatric comorbidity e.g. psychosis, severe depression, suicidality

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with Borderline personality disorder that are current in treatment in the inpatient dialectical behavioral therapy unit of the universityhospitel or have completed the treatment.
  Matched, healthy controls without psychiatric disorders
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Emotional reaction | one session of 90min
  Patients comparded to healthy controls will show a stronger emotional reaction on the stimuli.
  Patients more severely affected will show a stronger emotional reaction compared to less affected patients.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Philipsen, Prof., Principal Investigator — Department of Psychiatry and Psychotherapy - University Hospital, University of Oldenburg, Oldenburg, Germany
Locations (1):
- Department of Psychiatry and Psychotherapy - University Hospital, University of Oldenburg, Bad Zwischenahn, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bachmann K, Schulze M, Soros P, Schmahl C, Philipsen A. Development and validation of an emotional picture set of self-injury (EPSI) for borderline personality disorder: protocol for a validation study. BMJ Open. 2019 May 22;9(5):e027063. doi: 10.1136/bmjopen-2018-027063. PMID 31122985